CLINICAL TRIAL: NCT02760225
Title: 89Zr-pembrolizumab-PET Imaging in Patients With Locally Advanced or Metastatic Melanoma or Non-small Cell Lung Cancer
Brief Title: Pembrolizumab-PET Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201600163
Record Dates: First submitted 2016-03-29; First posted 2016-05-03 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Melanoma; Non-small Cell Lung Cancer
Keywords: Pembrolizumab; PET imaging; Melanoma; Non-small cell lung cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 89Zr-Pembrolizumab PET imaging (Experimental): In part A of the imaging trial, a dose finding imaging study will be performed to assess the optimal tracer protein dose of 89Zr-pembrolizumab and the optimal interval between tracer injection and scanning. Approximately 3 cohorts of about 2-3 patients each will undergo 89Zr-pembrolizumab-PET imaging before start of treatment with pembrolizumab. In part B, 12 eligible patients will undergo 89Zr-pembrolizumab-PET imaging at baseline, with the optimal tracer protein dose and scanning schedule as determined in part A.
  Interventions: Drug: 89Zr-Pembrolizumab; Device: 89Zr-Pembrolizumab PET

INTERVENTIONS:
Drug: 89Zr-Pembrolizumab — In part A of the imaging trial, a dose finding imaging study will be performed to assess the optimal tracer protein dose of 89Zr-pembrolizumab and the optimal interval between tracer injection and scanning. Approximately 3 cohorts of about 2-3 patients each will undergo 89Zr-pembrolizumab-PET imaging before start of treatment with pembrolizumab. In part B, 12 eligible patients will undergo 89Zr-pembrolizumab-PET imaging at baseline, with the optimal tracer protein dose and scanning schedule as determined in part A.
  Other Names: Injection of 89Zr-Pembrolizumab for imaging
Device: 89Zr-Pembrolizumab PET — In part A of the imaging trial, a dose finding imaging study will be performed to assess the optimal tracer protein dose of 89Zr-pembrolizumab and the optimal interval between tracer injection and scanning. Approximately 3 cohorts of about 2-3 patients each will undergo 89Zr-pembrolizumab-PET imaging before start of treatment with pembrolizumab. In part B, 12 eligible patients will undergo 89Zr-pembrolizumab-PET imaging at baseline, with the optimal tracer protein dose and scanning schedule as determined in part A.
  Other Names: 89Zr-Pembrolizumab PET scan(s)

SUMMARY:
This is a two center, single arm, investigator sponsored trial (IST) with the PET tracer 89Zr-pembrolizumab to evaluate in vivo whole body distribution of 89Zr-Pembrolizumab in a registered indication: locally advanced metastatic melanoma or non-small cell lung cancer before Pembrolizumab treatment.

DETAILED DESCRIPTION:
Rationale: Immunotherapy targeting specific immune-regulatory checkpoints, mainly cytotoxic T-lymphocyte antigen-4 (CTLA-4) and Programmed Death (PD1) or PD ligand 1 (PD-L1) have shown spectacular effects in a broad range of solid malignancies, including melanoma and non-small cell lung cancer (NSCLC). Pembrolizumab, is a monoclonal antibody that blocks the interaction between PD-1 on T-cells with its ligands PD-L1 and PD-L2. Anti-tumor activity with an acceptable side effect profile have been shown in melanoma and NSCLC.

Radio-labeling of pembrolizumab with the positron emission tomography (PET) radionuclide 89Zirkonium (89Zr) enables serial non-invasive imaging and quantification of distribution of PD-1 in melanoma patients. By performing a 89Zr-pembrolizumab-PET scan prior to treatment with pembrolizumab, the uptake of the tracer in the tumor lesions and normal organ distribution can be evaluated, this could lead to new insights about heterogeneity of PD-1 expression, as well as the use of a 89Zr-pembrolizumab-PET as a complementary tool for patient selection in the future.

Objective: Primary objective: To evaluate whole body distribution of 89Zr-pembrolizumab in patients with locally advanced or metastatic melanoma or NSCLC. Secondary objectives: i) To evaluate pharmacokinetics of 89Zr-pembrolizumab; ii) To assess the heterogeneity of 89Zr-pembrolizumab tumor uptake; iii) To describe safety of 89Zr-pembrolizumab; iv) To correlate the tumor response of pembrolizumab, as measured by objective response rate (ORR) according to standard RECIST v1.1 as assessed by the investigator, with specific tumor tracer uptake.

Study design: This is a two center, single arm, investigator sponsored trail (IST) with the PET tracer 89Zr-pembrolizumab to evaluate in vivo whole body distribution of 89Zr-pembrolizumab in a registered indication for locally advanced metastatic melanoma or NSCLC before Pembrolizumab treatment.

Study population: Eligible are patients with locally advanced or metastatic melanoma or NSCLC, who are eligible to receive Pembrolizumab treatment and who have at least one tumor site that is accessible for a tumor biopsy.

Intervention : In part A of the imaging trial, a dose finding imaging study will be performed to assess the optimal tracer protein dose of 89Zr-pembrolizumab and the optimal interval between tracer injection and scanning. Approximately 3 cohorts of about 2-3 patients each will undergo 89Zr-pembrolizumab-PET imaging before start of treatment with pembrolizumab. In part B, 12 eligible patients will undergo 89Zr-pembrolizumab-PET imaging at baseline, with the optimal tracer protein dose and scanning schedule as determined in part A. In total, a maximum of 21 patients will be included.The purpose of part B of the study is to analyze the whole body distribution and pharmacokinetics (PK) of 89Zr-Pembrolizumab. Tumor and normal organ radioactive tracer uptake will be quantified as standardized uptake values (SUV). Tumor biopsies will be collected at baseline and studied for various characteristics including Programmed cell death-ligand 1 (PDL-1), PD-1 expression and tumor infiltrating lymphocytes. Pembrolizumab treatment will be administered as standard of care Main study parameters/endpoints: To evaluate whole body distribution of 89Zr-pembrolizumab in patients with locally advanced or metastatic melanoma.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: For this imaging study patients have to make maximal 6 extra visits to the clinic for screening, to receive tracer injection and for maximal 3 PET/CT scans and the biopsy before start of standard treatment with pembrolizumab. The study ends after the last imaging or biopsy (whichever comes first) and will approximately take 7 days. Whenever possible, all procedures that are part of the study protocol will be planned during regular visits to the hospital as part of care as usual.

89Zr-pembrolizumab-PET/CT implements a radiation burden of about 20 millisievert (mSv), and 1.5 mSv per low-dose CT scan. Besides PET imaging, patients will be asked to give in total 12 blood samples (85 mL), which will give minor discomfort. A metastases biopsy will be performed, preferably from an easily accessible lesion to minimize the burden and risk for the patient. Based on a literature review, the risk of tumor biopsies is considered low with a small risk on significant/major complications or death. The risk associated with the 89Zr-pembrolizumab seems minor and although patients do not directly benefit from this study, results of this study will be valuable for our understanding of the tumor immune response and will guide further prospective research.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically documented locally advanced or metastatic melanoma or NSCLC.
3. Patients must be eligible for treatment with Pembrolizumab. For patients with NSCLC this includes PD-L1 expression (>1% based on IHC assay) on tumor material.
4. Metastatic lesion(s) (≥1,0 cm) of which a histological biopsy can safely be obtained according to standard clinical care procedures.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
6. Life expectancy ≥ 12 weeks .
7. Signed Informed Consent Form.
8. Ability to comply with protocol.
9. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions.
10. Adequate hematologic and end organ function, defined by the following laboratory results obtained within ≤ 14 days prior to 89Zr-pembrolizumab injection:

    * Absolute Neutrophil Count (ANC) ≥ 1500 cells/μL (without granulocyte colony-stimulating factor support within 2 weeks prior to 89Zr-pembrolizumab injection)
    * White Blood Count (WBC) ≥ 2500/μL
    * Lymphocyte count ≥ 500/μL
    * Platelet count ≥ 100,000/μL (without transfusion within 2 weeks prior to 89Zr-Pembrolizumab injection)
    * Hemoglobin ≥9.0 g/dL. Patients may be transfused or receive erythropoietin treatment to meet this criteria.
    * Asparate Aminotransferase (AST), Alanine Aminotransferase (ALT), and alkaline phosphatase ≤2.5 x the Upper Limit of Normal (ULN), with the following exceptions:

      * Patients with documented liver metastases: AST and/or ALT ≤ 5 x ULN
      * Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN
    * Serum bilirubin ≤ 1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level ≤3 x ULN may be enrolled.
    * International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (aPTT) ≤1.5 x ULN. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
    * Creatinine clearance ≥30 mL/min
11. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly).

Exclusion Criteria:

1. Any approved anti-cancer therapy, including chemotherapy of hormonal therapy within ≤14 days prior to 89Zr-pembrolizumab injection; the following exceptions are allowed:

   • Hormone-replacement therapy or oral contraceptives.
2. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to the 89Zr-pembrolizumab injection.
3. Malignancies other than melanoma or NSCLC within 5 years prior to 89Zr-pembrolizumab injection, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent or ductal carcinoma in situ treated surgically with curative intent).
4. Pregnant and lactating women.
5. Symptomatic brain metastasis.
6. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
7. Known hypersensitivity or allergy to any component of the pembrolizumab formulation.
8. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

   * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
   * Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
9. Positive test for Human Immunodeficiency Virus (HIV).
10. Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

    * Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to 89Zr-Pembrolizumab injection.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
11. Signs or symptoms of infection within 2 weeks prior to 89Zr-pembrolizumab injection.
12. Major surgical procedure other than for diagnosis within 28 days prior to 89Zr-pembrolizumab injection or anticipation of need for a major surgical procedure during the course of the study.
13. Prior allogeneic bone marrow transplantation or solid organ transplant.
14. Treatment with corticosteroids in an increasing dosage in the 7 days prior to 89Zr-pembrolizumab injection. (A stable or decreasing dosage of ≤ 1,5 mg dexamethasone or ≤ 10 mg prednisolone equivalent is allowed. In addition, inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease.)
15. Inability to comply with other requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Description of whole body 89Zr-pembrolizumab by measuring standardized uptake value (SUV) on the 89Zr-pembrolizumab-PET scans | 1 year

SECONDARY OUTCOMES:
Tumor and immune cell PD-L1 expression analysis in a fresh pre-treatment biopsy, and if available archival tumor biopsy, will be correlated to 89Zr-pembrolizumab tumor uptake, evaluated by measuring SUV on the 89Zr-pembrolizumab-PET. | 1 year
Safety assessment through summaries of adverse events, changes in laboratory test results, changes in vital signs, and exposure to 89Zr-pembrolizumab. Adverse event data will be recorded and summarized according to NCI CTCAE v4.0. | 1 year
  Safety assessment through summaries of adverse events, changes in laboratory test results (if evaluation is indicated), changes in vital signs, and exposure to 89Zr-pembrolizumab. Adverse event data will be recorded and summarized according to NCI CTCAE v4.0. Serious adverse events, including deaths, will be listed separately and will be summarized. For events of varying severity, the highest grade will be used in summaries. Relevant laboratory tests and vital signs (heart rate, respiratory rate, blood pressures, and temperature) data will be displayed by time, with Grade 3 and 4 values identified, where appropriate.
89Zr-pembrolizumab normal organ uptake on the 89Zr-pembrolizumab PET scans will be correlated to (89Zr-)pembrolizumab blood kinetics. | 1 year
  89Zr-pembrolizumab normal organ uptake on the 89Zr-pembrolizumab PET scans will be correlated to (89Zr-)pembrolizumab blood kinetics. Aliquots of whole blood and serum will be measured for 89Zr-activity in an isotope well counter and corrected for decay. Whole blood and serum activity will be expressed as standardized uptake value (SUV). Serum blood samples will also be collected regularly during the study to measure unlabeled pembrolizumab. PK parameters will be derived from the serum concentrations.
Evaluation of ORR according to standard RECIST v1,1 | 1 year
  Evaluation of ORR according to standard RECIST v1,1. ORR is defined as the proportion of subjects whose best overall response is either a PR or CR.

CONTACTS AND LOCATIONS:
Overall Officials: E. G.E. de Vries, Prof., Principal Investigator — Universit Medical Center Groningen
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen

REFERENCES:
- [Derived] Li W, Wang Y, Rubins D, Bennacef I, Holahan M, Haley H, Purcell M, Gantert L, Hseih S, Judo M, Seghezzi W, Zhang S, van der Veen EL, Lub-de Hooge MN, de Vries EGE, Evelhoch JL, Klimas M, Hostetler ED. PET/CT Imaging of 89Zr-N-sucDf-Pembrolizumab in Healthy Cynomolgus Monkeys. Mol Imaging Biol. 2021 Apr;23(2):250-259. doi: 10.1007/s11307-020-01558-w. Epub 2020 Oct 26. PMID 33104972